CLINICAL TRIAL: NCT03913234
Title: Phase IB & II Study of Ribociclib With Trastuzumab Plus Letrozole in Postmenopausal HR+, HER2+ Advanced Breast Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0765
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: HER2-positive Breast Cancer; Postmenopausal; Metastatic Breast Cancer
Keywords: HR-positive; HER2-positive; Breast Cancer; Hormone-positive; CDK4/6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Trastuzumab; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of Letrozole, Trastuzumab with Ribociclib (Experimental): Phase IB (dose escalation of ribociclib with fixed dose of letrozole and Ribociclib) Phase II (ribociclib of RPIID with fixed dose of letrozole and ribociclib)
  Interventions: Drug: Ribociclib, Trastuzumab, Letrozole

INTERVENTIONS:
Drug: Ribociclib, Trastuzumab, Letrozole — Phase IB: letrozole 2.5mg (fixed dose), trastuzumab (8mg/kg loading followed by 6mg/kg q 3weeks, fixed dose) plus ribociclib (dose escalation from 200mg to 600mg) to identify recommended phase iI dose (RPIID) Phase II: letrozole, trastuzumab (same as phase IB) plus ribocicilb RPIID

SUMMARY:
Survival benefit and quality of life are two key elements that should be kept in mind in the treatment of metastatic breast cancer. In this regards, endocrine therapy (ET) is strongly recommended in hormone receptor (HR) positive patients unless there is visceral crisis even though there is no concrete evidence that it is better than chemotherapy in terms of survival.

HER2 positive breast cancer is a subtype of breast cancer that showed the greatest improvement in terms of survival during the last decade due to trastuzumab based therapy. Recently, taxane and HER2 directed doublet including trastuzumab and pertuzumab (THP) is considered as standard of therapy based upon randomized phase 3 clinical trial (CLEOTATRA).

HER2 positive breast cancer can be divided into HER2 enriched subgroup (HR-HER2+) and luminal B subgroup (HR+HER2+) in biologic viewpoint because they are distinctly different subgroups in gene expression analysis. Accordingly, we are currently treating biologically different subtypes in a same way, which is CTx and anti-HER2 combination therapy (THP).

Luminal HER2+ subgroup has actually been tested with endocrine therapy (ET) and anti-HER2 therapy showed better PFS than ET alone (TAnDEM trial and trial comparing lapatinib plus letrozole versus letrozole alone) [2],[3] confirming existence of cross talk between ER and HER2 pathways in clinical setting. However, the combination regimen between ET and anti-HER2 therapy is not widely used in current practice in ER+HER2+ MBC patients because PFS seemed to be relatively shorter compared with chemotherapy based combination with anti-HER2 therapy even though several guidelines recommend it to be used as an initial treatment unless there is visceral crisis as they recommended ET alone first in ER+HER2- MBC (NCCN 2018).

Recently, various CDK4/6 inhibitors including palbociclib, abemaciclib, and ribociclib were approved by FDA based on the clinical trial results demonstrating prolonged PFS over ET alone when it was combined with ET in ER+ advanced breast cancer [4]. In PALOMA 2 biomarker study, it was beneficial regardless of ER and Ki67 expression status.

Reflecting quite durable PFS prolongation (10 month in PALOMA2) shown in ER+ disease (luminal A and luminal B subtype except HR+HER2+ patients) with CDK4/6 inhibitor on top of ET, the hypothesis of this trial is whether CDK4/6 inhibitor could prolong survival in luminal HER2 breast cancer as it did in ER+HER2-patients. In preclinical study, palbociclib showed activity in not only ER+ cell lines but also HER2 positive cell lines [5]. Also, in phase Ib trial, a CDK4/6 inhibitor from Lilly, abemaciclib showed acceptable toxicity with endocrine therapy or trastuzumab with response rate of around 20%.

Hence, as of today, it could be justified and warranted to conduct a prospective trial of ribocicib+letrozole+trastuzumab in order to take a look at its efficacy and toxicity in HR+HER2 + advanced breast cancer.

DETAILED DESCRIPTION:
This trial is performed in a multicenter, single-group, and phases IB and II clinical trial.

This is a single-group clinical trial of the effects of ribociclib, letrozole and trastuzumab in postmenopausal women with HR+, HER2+ advanced breast cancer. This trial consists of two parts. The first part is a phase IB study of increasing the dose of ribociclib from 200mg to 600mg in combination with letrozole 2.5mg and trastuzumab (8mg/kg followed by 6mg/kg every 3 weeks). In phase IB study, three to six patients will be enrolled for each dose group.

When the IB phase ends, patient enrollment will be discontinued for intermediate safety analysis, and after DLT analysis will determine recommended phase II phase II part will be started. The recommended phase II dose of ribocicib determined in phase IB part with ribociclib and trastuzumab (8mg/kg followed by 6mg/kg every 3 weeks) will be administered. Treatment is discontinued in the following cases.

* Progression of disease
* Uncontrolled toxicity
* Patient's death
* Withdrawal of consent In phase II part, 61 patients will be enrolled and the first 20 patients will be analyzed for run-in phase to confirm the safety of the therapy.

Regardless of treatment cycle, the disease will be evaluated in the same manner as the method used at the time of registration at intervals of 8 weeks for the first 18 months and at intervals of 12 weeks after that. If the progress of the disease is clinically suspected, additional tests can be performed

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥19 years
* Women with advanced (loco-regionally recurrent or metastatic) breast cancer not amenable for curative therapy
* Histologically and/or cytologically confirmed estrogen receptor positive and/or progesterone receptor positive breast cancer
* HER2 positive breast cancer (IHC 3+ or IHC 2+ and FISH, SISH or CISH+)
* Postmenopausal patient defined as either one of the following.

  * Prior bilateral ovariectomy
  * Age ≥ 60 years old
  * Age <60 years and amenorrhea over 12 months (without chemotherapy, tamoxifen, toremifene or ovarian inhibition), FSH and estradiol are in the postmenopausal range according to local normal range
* Patients who were not previously treated with systemic treatment for advanced / metastatic breast cancer
* ECOG performance status 0 or 1
* Measurable or evaluable lesion according to RECIST v1.1
* Normal organ function defined as

  * ANC (absolute neutrophil count) ≥ 1.5 × 109/L
  * Platelet ≥ 100 × 109/L
  * Serum Hb ≥ 9.0 g/dL
  * INR ≤1.5
  * Serum creatinine ≤ 1.5 X ULN
  * ALT & ALT < 2.5 X ULN (in the absence of liver metastasis) or ALT & ALT < 5 X ULN (with liver metastasis)
  * Total serum bilirubin < 1.5 X ULN
* Left Ventricular Ejection Fraction (LVEF) within normal range
* Voluntary agreement on clinical trials

Exclusion Criteria:

- Patients who have previously received CDK4 / 6 inhibitors or who have received other systemic treatments for advanced / metastatic breast cancer (Previous neo-adjuvant of adjuvant trastuzumab or aromatase inhibitor is not allowed, unless

1. Disease free interval was more than 12 months from the last dose of adjuvant trastuzumab or
2. Adjuvant aromatase inhibitor was administered more than 2 years)

   * Inflammatory breast cancer
   * Central nervous system metastasis
   * Active cardiac disease or a history of cardiac dysfunction including any of the following (Congestive heart failure within 6 months, history of myocardial infarction, unstable angina pectoris, or QTc prolongation on electrocardiogram)
   * Gastrointestinal absorption disorders that interfere with drug absorption
   * Patients who is currently receiving medications that can prolong QT intervals (QTc>450msec) on ECG or that can cause torsades de pointes
   * Patients with severe visceral metastasis on enrolment who are not indicated with hormone treatment
   * Serious surgical treatment within 14 days prior to study treatment
   * Radiotherapy within 21 days prior to study treatment
   * Serious medical comorbidities
   * Concurrent malignancy or malignancy within 3 years of study participation, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 95 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 1 year
  Progression free survival is defined as the time from the start of investigational drug to disease progression or patient's death whichever occurred first

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival is the time from the start of investigational drug to patient's death.
Response rate | 1 year
  Response rate is defined as the response to the drug according to RECIST v1.1 criteria.
Quality of life | 1 year
  Overall survival is the time from the start of investigational drug to patient's death Response rate is defined as the response to the drug according to RECIST v1.1 criteria Quality of life will be measured using EORTC-QLQ C30 questionaire. (Purpose of EORTC-QLQ C30 is to measure the quality of life of the subjects who participated in the clinical study. It consists of 30 questions and each question will be answered by 4 scale answers "Not at all", "A little", "Quite a bit", and "Very much".)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center at Yonsei University Health System, Seoul, South Korea